CLINICAL TRIAL: NCT01133704
Title: A Randomized, Double Blind, Placebo Controlled Trial of Immunotherapy With Autologous Antigen-Loaded Dendritic Cells (Provenge®, APC8015) for Asymptomatic, Metastatic, Hormone-Refractory Prostate Cancer
Brief Title: Immunotherapy With APC8015 (Sipuleucel-T, Provenge) for Asymptomatic, Metastatic, Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dendreon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9902A
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Hormone-Refractory Prostate Cancer
Keywords: asymptomatic metastatic hormone-refractory prostate cancer
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- sipuleucel-T (APC8015) (Active Comparator)
  Interventions: Biological: sipuleucel-T
- Placebo (Placebo Comparator)
  Interventions: Biological: APC-Placebo

INTERVENTIONS:
Biological: sipuleucel-T
  Arms: sipuleucel-T (APC8015)
Biological: APC-Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled trial of immunotherapy with autologous antigen-loaded dendritic cells (Provenge, APC8015) for asymptomatic, metastatic, hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Metastatic disease as evidenced by soft tissue and/or bony metastases
* Prostate-specific antigen value of at least 5 ng/mL
* Tumor progression while on hormonal therapy
* Castration levels of testosterone (defined as less than 50 ng/dL)
* Life expectancy of at least 16 weeks
* Adequate hematologic, renal, and liver function

Exclusion Criteria:

* Visceral organ metastases
* Metastatic disease expected to be in need of radiation therapy within 4 months.
* Concurrent therapy with experimental agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2000-05; Primary Completion 2003-03 (Actual); Study Completion 2005-05 (Actual)

REFERENCES:
- [Derived] Ju M, Fan J, Zou Y, Yu M, Jiang L, Wei Q, Bi J, Hu B, Guan Q, Song X, Dong M, Wang L, Yu L, Wang Y, Kang H, Xin W, Zhao L. Computational Recognition of a Regulatory T-cell-specific Signature With Potential Implications in Prognosis, Immunotherapy, and Therapeutic Resistance of Prostate Cancer. Front Immunol. 2022 Jun 23;13:807840. doi: 10.3389/fimmu.2022.807840. eCollection 2022. PMID 35812443
- [Derived] Small EJ, Higano CS, Kantoff PW, Whitmore JB, Frohlich MW, Petrylak DP. Time to disease-related pain and first opioid use in patients with metastatic castration-resistant prostate cancer treated with sipuleucel-T. Prostate Cancer Prostatic Dis. 2014 Sep;17(3):259-64. doi: 10.1038/pcan.2014.21. Epub 2014 Jun 24. PMID 24957547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between May 2000 and March 2003 across 24 clinical trial sites.
Pre-assignment Details: Participants were screened for evaluation of subject eligibility and performance of baseline tests/procedures.
Groups:
- Sipuleucel-T (APC8015): All subjects randomized to receive sipuleucel-T.
  Autologous peripheral blood mononuclear cells, including antigen presenting cells, that have been activated in vitro with a recombinant fusion protein, PAP-GM-CSF. Treatment consist of 3 doses administered approximately 2 weeks apart.
- Placebo: All subjects randomized to receive placebo.
  Approximately one-third of the autologous quiescent APCs prepared from a single leukapheresis procedure. A course of therapy consists of 3 complete doses given at approximately 2-week intervals.
Period: Overall Study
Arm/Group | Sipuleucel-T (APC8015) | Placebo
Started | 65 | 33
Completed | 16 ((including 3 year follow-up)) | 7 ((including 3 year follow-up))
Not Completed | 49 | 26
Not completed — Death | 44 | 26
Not completed — Patient refused to continue | 4 | 0
Not completed — Study Closure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sipuleucel-T (APC8015) | Placebo | Total
Number analyzed (Participants) | 65 | 33 | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.2) | 70.6 (7.8) | 69.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 65 | 33 | 98

OUTCOME MEASURES:

1. Primary Outcome: Overall Time to Disease Progression
Description: Overall time to disease progression in subjects with asymptomatic metastatic hormone-refractory prostate cancer treated with sipuleucel-T (APC8015) compared to overall time to disease progression in subjects treated with placebo.
Time Frame: from randomization to 36 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sipuleucel-T (APC8015) | Placebo
Number analyzed (Participants) | 65 | 33
Weeks | 10.9 [9.3 to 17.7] | 9.9 [8.4 to 18.0]
Statistical Analysis 1: Comparison: Sipuleucel-T (APC8015) vs Placebo; Test type: Superiority or Other; p = 0.719, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.69 to 1.70] — Obtained from a Cox proportional hazards model with treatment group as the independent variable, stratified by bisphosphonate use (placebo/sipuleucel-T)

2. Secondary Outcome: Overall Survival
Description: Subjects were followed for 3 years from the time of randomization or until death.
Time Frame: Time from randomization until 36 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sipuleucel-T (APC8015) | Placebo
Number analyzed (Participants) | 65 | 33
Months | 19.0 [13.6 to 31.9] | 15.7 [12.8 to 25.4]
Statistical Analysis 1: Comparison: Sipuleucel-T (APC8015) vs Placebo; Test type: Superiority or Other; p = 0.331, Log Rank; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.78 to 2.07] — Obtained from a Cox proportional hazards model with treatment as the independent variable, and stratified by bisphosphonate use (placebo/sipuleucel-T)

ADVERSE EVENTS:
Time Frame: From randomization through 36 months. Median follow-up was 36 months.
Description: Safety population: All subjects randomized to each arm who underwent at least one leukapheresis procedure. Not all randomized subjects underwent at least one leukapheresis procedure.
Arm/Group | Sipuleucel-T (APC8015) | Placebo
Serious Adverse Events (participants affected / at risk) | 13/65 | 9/31
Other Adverse Events (participants affected / at risk) | 63/65 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (APC8015) (N=65) | Placebo (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Chills (General disorders) | 3 | 0
Disease Progression (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain mass (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sipuleucel-T (APC8015) (N=65) | Placebo (N=31)
Anaemia (Blood and lymphatic system disorders) | 13 | 1
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Hypoaesthesia Oral (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1
Asthenia (General disorders) | 12 | 2
Chills (General disorders) | 34 | 2
Fatigue (General disorders) | 27 | 5
Influenza Like Illness (General disorders) | 4 | 2
Malaise (General disorders) | 4 | 0
Oedema Peripheral (General disorders) | 7 | 5
Pain (General disorders) | 9 | 2
Pyrexia (General disorders) | 19 | 3
Citrate Toxicity (Injury, poisoning and procedural complications) | 10 | 5
Anorexia (Metabolism and nutrition disorders) | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 7
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 8 | 2
Headache (Nervous system disorders) | 14 | 3
Lethargy (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 6 | 5
Paraesthesia Oral (Nervous system disorders) | 5 | 3
Tremor (Nervous system disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 1 | 4
Urinary Retention (Renal and urinary disorders) | 3 | 2
Gynaecomastia (Reproductive system and breast disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 0
Pallor (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A provision provides for sponsor review up to 45 days with the right to request modification based on disclosure of confidential information; extendable by 60 days to file a patent application.